CLINICAL TRIAL: NCT06619184
Title: Comparison of The Effectiveness Between Transplantation of Autologous Non-Cultured Extracted Hair Follicle Outer Root Sheath Cell Suspension and Mini Punch Graft in Non-Segmental Vitiligo
Brief Title: Transplantation of Autologous Non-Cultured Extracted Hair Follicle Outer Root Sheath Cell Suspension and Mini Punch Graft for Stable Non-Segmental Vitiligo Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DV-202407.01.
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Non Segmental Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCEHFORSCS transplantation and MPG procedure (Experimental): The research was conducted on 21 participants.
  Two vitiligo lesions from each participant that met the inclusion and exclusion criteria were treated with NCEHFORSCS transplantation and MPG procedure followed by observation of repigmentation.
  The participants were informed that a series of procedures would be performed, including hair follicle extraction using the follicle unit extraction (FUE) procedure, followed by the preparation of NCEHFORSCS in PT Prodia StemCell Indonesia (ProSTEM®) laboratory, and transplantation of NCEHFORSCS on one VNS lesion while MPG procedure was performed on another lesion.
  Follow-up was carried out at the 2nd week, 4th week, 8th week, 12th week, and 16th week after the NCEHFORSCS transplantation and MPG procedures to assess repigmentation of the lesions and side effects of the procedures.
  Interventions: Procedure: NCEHFORSCS transplantation; Procedure: MPG procedure

INTERVENTIONS:
Procedure: NCEHFORSCS transplantation — One vitiligo lesion of participans treated with NCEHFORSCS transplantation including follicle unit extraction (FUE) procedure from the occipital area, laboratory procedure for preparation of cell suspension, and transplantation of NCEHFORSCS.
Procedure: MPG procedure — Another vitiligo lesion treated with MPG procedure
  Follow up The dressing was removed by the researcher on day 8 The participants were asked to attend for follow-up at the clinic on week 2, 4, 8, 12, and 16 after the two procedure were done.
  At 2, 4, 8, 12 and 16 weeks of follow-up visits, any possible complications were evaluated and digital photographs of the lesions were taken for evaluating the two procedure efficacy using its parameter: appearance of repigmentation (AOR), total number of repigmentation NSV lesions, extent area of repigmentation, and color match

SUMMARY:
Vitiligo is an acquired pigmentation disorder due to loss of melanocytes characterized by depigmentation macules or patches. One type of this disease is nonsegmental vitiligo (NSV). Until now, there is no satisfactory treatment for vitiligo. Vitiligo therapies are medical therapy include topical and systemic therapy, phototherapy as well as surgery. Surgical treatment is indicated in stable vitiligo, which is not responding to medical treatment. This procedure consists of tissue grafting and cellular transplantation. Mini punch graft (MPG) is the most frequently performed tissue transplantation technique, while cellular transplantation from autologous noncultured extracted hair follicle outer root sheath cell suspension (NCEHFORSCS) containing melanocyte stem cells, is currently a promising option.

DETAILED DESCRIPTION:
Current NSV treatments can be considered suboptimal and leading to decreased patient's quality of life due to the emotional burden of therapy dissatisfaction. When a stable NSV is not responding to medical therapy, surgery may be a useful treatment approach. All surgical techniques in vitiligo treatment share the same principle: transferring autologous melanocytes from a donor to repopulate melanocytes in the depigmented area that lacks a reservoir or fails to activate melanocytes in the outer root sheath (ORS) of hair follicles. MPG as the most frequently performed tissue transplantation technique transferred the epidermal melanocyte to vitiligo lesion, while NCEHFORSCS provides melanocytes with better properties and contains melanocyte stem cells. The advantages of melanocytes from ORS compared to epidermal are the follicular melanocyte:keratinocyte ratio consists of one melanocyte for every five keratinocytes or 1:5 in the hair bulb, melanocytes are more dendritic, have larger melanosomes, and have the potential to produce more melanin pigment. Due to these properties, hair follicles can be a better source of melanocytes than epidermis in the delivery of cellular transplantation-based therapy for vitiligo therapy. Research comparing the effectiveness of the two procedures has never been conducted in Indonesia, even though the incidence of vitiligo is quite high and the success of therapy is still not optimal. So the purpose of this study is to compare the effectiveness of the two procedures in NSV patient.

ELIGIBILITY:
Inclusion Criteria:

1. Non-Segmental Vitiligo patients
2. Minimal 1-year duration of stability
3. Age between 18-70 years
4. Having at least two vitiligo lesions for NCEHFORSCS transplantation and MPG procedure

The two vitiligo lesions to be treated must meet the following criteria:

1. Have similar size, minimum of 1 cm² and a maximum of 20 cm²
2. The distance between the two lesions at least 1 cm
3. Location of the lesions must have a relatively similar distribution of hair follicles
4. Not located on the palms, soles, or penis

Exclusion Criteria:

1. Pregnant
2. Active vitiligo
3. Mixed vitiligo
4. Presence of new lesions
5. History of hypertrophic scars and keloids
6. History of bleeding disorders
7. Other active autoimmune diseases
8. History of wound healing disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Appearance of repigmentation (AOR) | 4 months
  The first appearance of repigmentation in non-segmental vitiligo (NSV) lesions after NCEHFORSCS transplantation and MPG procedure evaluated by blind investigator using dermoscope at weeks 2, -4, -8, -12, and -16
Total number of repigmentation non-segmental vitiligo (NSV) lesions | 4 months
  Total number of NSV lesions that experienced repigmentation at the 16th week of observation
Extent area of repigmentation | 4 months
  The repigmentation area percentage level of non-segmental vitiligo (NSV) lesions after NCEHFORSCS transplantation and MPG procedure determine by blind investigator using the digital images.
  The scores were confirmed by objective measurement of the extent of repigmentation by a digital image analysis system ImageJ® as follow:
  No repigmentation (0%) Poor repigmentation (0,1-49%) Fair repigmentation (50-74%) Good repigmentation (75-89%) Excellent repigmentation (90-100%)
Color match | 4 months
  Color match between repigmentation of the lesions and surrounding skin assessed subjectively by a blind investigator using digital photography at week 16 as follows:
  No repigmentation color Lighter than peri lesion skin color Same as peri lesion skin color Darker than peri lesion skin color

SECONDARY OUTCOMES:
Complication | 4 months
  Complication at the location of melanocyte donor and recipient both from the two procedure include secondary infection, milia, scar tissue, rejection, and new vitiligo lesion (Köebnerization) on the donor or recipient site of NCEHFORSCS transplantation and cobblestone appearance at the recipient area of MPG and minimal superficial scar tissue at the MPG donor area.

CONTACTS AND LOCATIONS:
Overall Officials: Reiva Farah Dwiyana, MD, Principal Investigator — Universitas Padjadjaran
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia